CLINICAL TRIAL: NCT06771791
Title: Evaluation of the Efficacy of Oral Immunotherapy with Raw Apple in Patients Allergic to Birch Pollen and Apple: Prospective, Multicenter, Comparative Phase III Study
Acronym: ELIO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9432
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Allergies
Keywords: allergy; oral immunotherapy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral immunotherapy (Experimental): oral immunotherapy with raw apple during 9 month
  Interventions: Other: oral provocation test
- eviction (Placebo Comparator): avoidance of raw apples for 9 months
  Interventions: Other: oral provocation test

INTERVENTIONS:
Other: oral provocation test — Progressively increasing doses of peeled fresh Golden apple or placebo will be consumed by the patient (4g, 12g, 40g, 120g) with a time interval of 20 minutes between each dose.

SUMMARY:
Apple-birch pollen-food allergy syndrome is particularly common in Northern and Central Europe (70% of patients allergic to birch pollen), and classically induces an oral syndrome that impairs patients' quality of life. Current treatment is based on food avoidance. However, evidence of the efficacy of this treatment is limited (small numbers, lack of validation with a control group, absence of double-blind evaluation of the primary endpoint in a challenge test against placebo). The aim of oral immunotherapy with raw apple is to improve the management of allergic patients by enabling them to acquire tolerance to raw apple and other rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Patient with allergic rhinitis to birch pollen.
* Patient with an oral syndrome within 15 minutes of consuming at least one of the first 3 doses of raw apple in the V0 or V1 raw apple oral challenge test.
* Evidence of sensitization to PR10 proteins in birch pollen and apple: positive prick tests to birch pollen and raw Golden apple and/or positive Bet v 1 and Mal d 1 specific IgE assays.
* Subject affiliated to a social health insurance scheme
* Subject able to understand the aims and risks of the research and to give dated and signed informed consent
* For women of childbearing age: negative urine pregnancy test at inclusion visit

Exclusion Criteria:

* Severe or uncontrolled asthma
* Severe obstructive syndrome
* Active neoplastic disease
* Active autoimmune disease
* Eosinophilic esophagitis or other active eosinophilic gastrointestinal pathologies
* History of bariatric surgery
* History of anaphylaxis to apples
* Allergy to cooked apples
* Contraindication to anti-histamines, corticoids, salbutamol, adrenaline
* Other contraindication to an oral challenge test
* Allergy to placebo ingredients
* Presence of oral syndrome during consumption of placebo in the first oral challenge test
* Allergenic immunotherapy to birch pollen in progress or completed less than 5 years ago
* Current treatment with anti-IgE, anti-IL4/13, anti-IL5 or anti-TSLP biotherapy.
* Impossibility of giving the subject informed information
* Subject under court protection
* Subject under guardianship or curatorship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of oral immunotherapy to raw apple on the reduction of oral raw apple syndrome | 9 month
  To evaluate the efficacy of oral immunotherapy to raw apple on the reduction of oral raw apple syndrome after 9 months of oral immunotherapy. A reduction in oral syndrome after 9 months of oral immunotherapy with raw apple is defined as: absence of oral syndrome on the 9-month raw apple OPT when consuming a dose of raw apple 3 times greater than the dose of raw apple triggering oral syndrome on the initial raw apple oral challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France, France

IPD SHARING:
Plan to Share IPD: Undecided